CLINICAL TRIAL: NCT06231407
Title: Recovery Oriented Cognitive Therapy (CT-R) Medication Checks: An Acceptability and Feasibility Trial, Standard Operating Procedure
Brief Title: Increasing Medication Check Participation Through Applying CT-r
Acronym: IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Aaron Brinen, Assistant Professor of Psychiatry and Behavioral Sciences, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 220048
Record Dates: First submitted 2023-07-19; First posted 2024-01-30 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Schizophrenia and Related Disorders
Keywords: Schizophrenia Spectrum Diagnosis; Cognitive Therapy; Cognitive Behavioral Therapy for Psychosis (CBTp); Recovery-Oriented Cognitive Behavioral Therapy for Psychosis; CT-R; Medication Management Appointments
MeSH Terms: conditions — Schizophrenia | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Subjects were recruited from an existing psychosis clinic and assigned to the participating psychiatry resident. A small group were misaligned and reconnected to use their data as a comparison for someone not receiving the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recovery Oriented CBTp Med Check (Experimental): Resident physicians will provide medication appointments, supervised by their attending physician (Stovall) and CT-R supervisor (Brinen). They will conduct their appointment per protocol detailed in a treatment manual. No additional/special information needs to be recorded in medical record, beyond the clinical notes expected per VAPOC policy. Appointments will be a standard length.
  Interventions: Behavioral: Recovery Oriented CBTp Medication Management
- Treatment as Usual (Active Comparator): Patient will attend traditional medication management check appointments with psychiatry residents.
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Recovery Oriented CBTp Medication Management — The prescriber structures the medication appointment to elicit and focus on subjects long term, valued goals (aspirations). With this information the prescriber will develop a plan to increase daily activity to facilitate the aspiration's pursuit. Obstacles (psychotic symptoms, motivational problems) will be identified and a formulation developed with the individual. Psychosocial interventions will be implemented for the various obstacles alongside monitoring and implementing of medications. Across sessions, the prescriber will continue to implement and monitor psychosocial interventions.
  Other Names: Recovery Oriented Cognitive Therapy
  Arms: Recovery Oriented CBTp Med Check
Behavioral: Treatment as Usual — Residents will conduct medication management appointments as normally conducted
  Other Names: TAU
  Arms: Treatment as Usual

SUMMARY:
The goal of this feasibility and acceptability trial is to learn about the acceptability of adding a recovery-oriented, psychological framework to a standard medication management appointment with a psychiatrist and any impact on attendance and functioning. The main question[s] it aims to answer are:

1. Will CT-R medication checks will be acceptable to the patient and feasible to deliver and receive, as measured by asking patients how they like the CT-R med checks and our ability to do this study in addition to number of patient drop-outs?
2. Will CT-R medication checks will be related to significantly greater engagement with treatment as measured by: lower no-show rates, greater self-reported working alliance, and better treatment adherence?
3. Will CT-R medication checks will be related to greater activity and increase in functioning as measured by: time use survey, GAF, skill use?
4. Will CT-R medication checks will be related to a trend in improved defeatist beliefs, negative symptoms, paranoia, and self-esteem?

Researchers will compare the group assigned to the trial psychiatrists to a small group who were assigned to non-trial psychiatrists to see if the intervention impacted any of the above questions beyond TAU.

DETAILED DESCRIPTION:
The current study aims to test whether adapting a psychological treatment for schizophrenia to medication appointments with psychiatry residents is acceptable and feasible, and whether it improves treatment engagement, functioning and symptom burden, particularly negative symptoms. In addition to providing psychiatry residents with a framework for conducting medication appointments, it will also give patients with psychotic disorders access to empirically-supported psychological interventions, that they may not otherwise have access to. We will test the acceptability and feasibility of this adapted intervention and examine whether effect sizes of change with intervention in this sample size warrant testing in a larger study.

Only patients who consent to being in the study will receive CT-R medication appointments. CT-R is a therapy process that is being implemented within the medication appointments. The provided measures and tasks are outcomes to be measured throughout the study. For instance, we are interested in how clinical symptoms, subjective well-being, and treatment engagement change with the implementation of CT-R in medication appointments.

1. CT-R medication checks will be acceptable to the patient and feasible to deliver and receive, as measured by asking patients how they like the CT-R med checks and our ability to do this study in addition to number of patient drop-outs.
2. CT-R medication checks will be related to significantly greater engagement with treatment as measured by: lower no-show rates, greater self-reported working alliance, and better treatment adherence
3. CT-R medication checks will be related to greater activity and increase in functioning as measured by: time use survey, GAF, skill use
4. CT-R medication checks will be related to a trend in improved defeatist beliefs, negative symptoms, paranoia, and self-esteem
5. Exploratory analyses will include:

   1. CT-R med checks will be related to greater improvement on a cognitive motivation task (EEfRT/Balloon task)
   2. Improvement in Defeatist Belief Scale (DBS) and Neg Symptoms will be mediated by increased treatment adherence, engagement and activity

Expected study duration: 3 years

3. Procedures_________________________________________________________________

4.1 Recruitment Vanderbilt Adult Psychiatry Outpatient Clinic (VAPOC): Individuals who are currently being seen for medication management through VAPOC, and who meet eligibility criteria, will be identified by the treating providers and study staff through review of medical records and consultation with providing clinicians. Potential participants will only be approached with the approval of the treating provider, who will determine whether that individual is likely to have the capacity to consider the research study and provide consent. If appropriate, their provider will ensure that the patient is agreeable to being approached about a research study or introduce the patient to the research team. Potential participants will be approached by research staff after their appointment for a brief screening visit.

Recruitment may occur in person, over telehealth, or over the phone. VAPOC accommodates both in-person and telehealth appointments, depending on the patient's preference. Therefore, for eligible patients who are seen regularly over telehealth, recruitment may occur by joining the telehealth appointment at the end of the visit. Additionally, potential participants may not be available to stay after their appointment, despite interest in the study. Therefore, individuals identified as a good fit, who cannot be connected with in-person, will be called on the phone for a screening, with the provider's consent and after the provider has ensured that the patient is agreeable to being called about a research study.

Resident subjects will be recruited from Vanderbilt Adult Psychiatry Outpatient Clinic. Residents who are involved with the study will be contacted either by email or in-person to assess their interest in being enrolled and consented as a participant in order for the research team to gather information about the acceptability and feasibility of carrying out the intervention.

4.3 Planned enrollment: We plan to recruit up to 40 subjects for the study.

4.4 Screening and Consent: Potential research subjects will be asked if they would like to participate in the current study. If they report potential interest, a pre-screening will occur. This screening will occur in person, over the phone or over telehealth (Zoom) using the Screening Form or Phone Script. Informed consent will be obtained by study personnel directly involved in the research (i.e. research staff or PI). Personnel have completed IRB training and have considerable experience running studies in clinical populations.

Informed consent will be obtained either, 1) in the research offices at the Psychiatric Neuroimaging Program or 2) over Zoom during a virtual study visit. A research staff member will explain the applicable procedures and the possible risks and benefits to the subjects. The details of the informed consent procedure are as follows:

1. The investigator or research staff and the subject will read together the entire consent form.
2. The subject will be asked details about the study. To document that the subject has read the consent form and has the capacity to understand the most important details, the investigator will use the appropriate Informed Consent Survey. The questions will be read by the investigator or research staff and the answers will be recorded. If the subject is unable to answer any of the questions, or if the subject demonstrates a lack of understanding, the investigator or research staff member will then review the details of the study again. Subjects who are unable to answer the questions, even after additional information is provided, will be excluded from the study.
3. The subject will be informed that regardless of whether or not they take part in this research study, it will not affect their treatment, payment or enrollment in any health plans or affect their ability to get benefits or care in any way.
4. The subject will be provided with copies of the signed consent form and the Informed Consent Survey (including the answers given) at the time of the initial visit. If completed virtually, this will be emailed, using secure email methods, to the subject with their consent.
5. At each visit, we will 1) remind participants that the research visit is voluntary (no matter how many previous visits they have done) and 2) ask them to tell us what they believe the purpose of the study is and repeat back what they will be doing that day (e.g. cognitive tasks, self-reports).

It will be emphasized to all subjects that their participation is completely voluntary, and that even after signing the consent document they are still free to withdraw from the study at any time. It will also be emphasized that if they choose to leave the study, their medication management at VAPOC will not be impacted, and they can continue seeing their medication provider as usual.

4.5 Intervention Assignment

Participants will not be randomized. Instead, they will serve as their own controls. Individuals will be recruited during Spring 2022 as described in section 3.1. Following their baseline assessment, participants will continue treatment as usual (TAU) with their current provider. The amount of time they are in the TAU branch of the study will depend on their date of recruitment. The intervention phase of the study will occur between August 2022- June 2023, after the patient has established care with their new provider. Therefore, a participant who was recruited in April 2021 may have a TAU duration of 5 months, whereas a participant who was recruited in June 2021 may only have TAU of 2 months. Participants not assigned to a resident associated with the study will continue in the study as controls, given their re-consent.

4.7 Medication appointments

Resident physicians will provide medication appointments, supervised by their attending physician (Stovall) and CT-R supervisor (Brinen). They will conduct their appointment per protocol (see below). No additional/special information needs to be recorded in medical record, beyond the clinical notes expected per VAPOC policy. Appointments will be a standard length.

No-shows and hospitalizations will be recorded in the chart per clinic procedures and will be monitored and recorded by study staff, with additional support from the Informatics team.

4.8 Video/Audio Recording

In order to ensure treatment fidelity, medication appointments will be video and/or audio recorded. Further, the qualitative interviews will be audio-recorded for later analyses. All recordings will be included in the Informed Consent document and described to the participants prior to study enrollment. Physicians will upload their sessions to a folder on Vanderbilt University Medical Center (VUMC) Box, which will only be available to necessary study staff for review. Additionally, qualitative interview recordings will be uploaded to a folder on VUMC Box, which will only be available to necessary study staff for review.

ELIGIBILITY:
Inclusion Criteria:

1. 18-80 years old
2. Schizophrenia-spectrum disorder
3. Typically scheduled 1x/month
4. Willingness to complete 2-3 hours of testing at multiple timepoints
5. Likely to stay in our clinic for the next 1-2 years

Exclusion Criteria:

1. Significant intellectual disability
2. Autism spectrum disorder
3. Cannot read/write English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-12-06 (Actual)

PRIMARY OUTCOMES:
Working Alliance Inventory | Upon Enrollment in the study, Up to 4 months later, At study completion (average of 1 year)
  Measure of patient perception of working alliance
Time Use Interview | Upon Enrollment in the study, Up to 4 months later, At study completion (average of 1 year)
  Interview capturing amount of time in productive activity.
Mental Illness Research Education and Clinical Center (MIRECC) Global Assessment of Functioning (GAF) | Upon Enrollment in the study, Up to 4 months later, At study completion (average of 1 year)
  Standardized Measure of overall functioning; Scored from 0-100 with higher score indicating better functioning. Scoring is based on predetermined parameters.
Compass | Upon Enrollment in the study, Up to 4 months later, At study completion (average of 1 year)
  Interview of symptoms and their severity.

SECONDARY OUTCOMES:
Defeatist Beliefs Scale | Upon Enrollment in the Study, on average the first of the month until the final assessment (approximately 15 months)
  Belief scale; 5 item scale rating agreement with a statement from 1 (Totally Agree) to 7 (Disagree Totally); Higher score indicates fewer defeatist beliefs. Minimum Value: 5, Maximum Value: 35
Asocial Beliefs Scale | Upon Enrollment in the Study, on average the first of the month until the final assessment (approximately 15 months)
  Belief scale; 7 item yes-no self-report questionnaire asking about one's interaction with others; Minimum Value: 7, Maximum: 14; Higher score indicates more beliefs about not socializing.
Cognitive Insight Scale | Upon Enrollment in the Study, on average the first of the month until the final assessment (approximately 15 months)
  Belief scale: Related to various forms of insight; 15-item self-report questionnaire designed to evaluate patients' self-reflectiveness and their overconfidence in their interpretations of their experiences. The scale demonstrates good convergent, discriminant, and construct validity; Statements are rated on a 4 point scale from 1-4 (Do Not agree at all; Agree completely); 6 of the items (2, 7, 9, 10, 11, 13) are reverse scored; Minimum Value: 15, Maximum Value: 60 Higher score indicates better cognitive insight.
Green Paranoid Thoughts Scale | Upon Enrollment in the Study, on average the first of the month until the final assessment (approximately 15 months)
  Thought scale of paranoia. 32 item assessment designed to evaluate patients' paranoia in social and interpersonal situations. Minimum Value: 32 Maximum Value is 160; Higher score indicating worse paranoia.
Self Esteem Scale | Upon Enrollment in the Study, on average the first of the month until the final assessment (approximately 15 months)
  Measure of individuals self esteem. is a 38 item self-reported questionnaire designed to measure the self and perceived self- esteem. Minimum Value: 38 Maximum Value is 380. Lower value indicates lower self esteem.
SOLES | Upon Enrollment in the Study, on average the first of the month until the final assessment (approximately 15 months)
  16 item (rated 0-10 agreement with statement) measurement of beliefs about mental health treatment and problems. Lower score is worse and higher score is better beliefs about mental health treatment. Minimum Value: 0, Maximum Value: 160
Questionnaire about the Process of Recovery (QPR) | Upon Enrollment in the Study, on average the first of the month until the final assessment (approximately 15 months)
  Measure of Recovery; 17 item questionnaire that measures the process of recovery. Each statement is rated regarding agreement on a 1-5 scale ranging from Disagree Strongly to Agree Strongly. Lower scores are indicative of worse beliefs about recovery. Minimum Value: 17, Maximum Value: 85

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Grant PM, Huh GA, Perivoliotis D, Stolar NM, Beck AT. Randomized trial to evaluate the efficacy of cognitive therapy for low-functioning patients with schizophrenia. Arch Gen Psychiatry. 2012 Feb;69(2):121-7. doi: 10.1001/archgenpsychiatry.2011.129. Epub 2011 Oct 3. PMID 21969420